CLINICAL TRIAL: NCT04192643
Title: THE IMPACT OF TRANEXAMIC ACID USAGE DURING LAPAROSCOPIC MYOMECTOMY
Brief Title: INTERVENTION WITH TRANEXAMIC ACID TO REDUCE HAEMORRHAGE DURING LAPAROSCOPIC MYOMECTOMY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alkü Alanya Education and Research Hospital (Other)
Responsible Party: Principal Investigator, MERAL TUĞBA ÇİMŞİR, ASSOCIATE PROFESSOR, Alkü Alanya Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: ALKU EDUCATION AND RESEARCH
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Uterine Fibroid; Myoma;Uterus; Tranexamic Acid Adverse Reaction
Keywords: uterin fibroid, laparoscopic myomectomy
MeSH Terms: conditions — Leiomyoma; Myofibroma | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: PROSPECTİVELY DOUBLE-BLİND RANDOMİSED CONTROLLED TRİAL
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TRANEXAMİC ACİD (Experimental): . 1 gr tranexamic acid in 100 ml salin given in 15 minutes
  Interventions: Drug: Tranexamic Acid 100 MG/ML
- NO TRANEXAMİC ACİD (Placebo Comparator): 100 ml salin solution
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Tranexamic Acid 100 MG/ML — 1 GR TRANEXAMİC ACİD İN 100 ML SALİNE SOLUTİON GİVEN İN 15 MİNUTES
  Arms: TRANEXAMİC ACİD
Drug: Placebos — 100 ML SALİNE SOLUTİON
  Arms: NO TRANEXAMİC ACİD

SUMMARY:
This research is planned as a randomised double-blind controlled trial. interventions to reduce haemorrhage during laparoscopic myomectomy for fiboids is important. İntraoperative Tranexamic acid usage can reduce haemorrhage and related symptoms when given during laparoscopic myomectomy. There is no randomised controlled trials in literature about tranexamic acid usage in laparoscopic gynecological operations.

DETAILED DESCRIPTION:
researchers planned this trial by firstly randomising the patients. 1 gr tranexamic acid in 100 ml salin will bi given by initial of the anesthesia of the patient, the other group will be taken only 100ml saline solution. Randomising will be double blind and only anesthesiologist will see if the paient is in working group or control group. Than researchers provide laparoscopic myomectomy with same prothocol to each patient. At the end of the operation, researchers will record all the parameters during operation like; operation starting and ending time, the amount of bleeding, time of suturing, the size, location and count of myoma uteri, complications, weight of myoma uteri and the change of haemoglobine levels before and after operation.

ELIGIBILITY:
Inclusion Criteria:

* myoma uteri
* appropiate for laparoscopy

Exclusion Criteria:

* malignancy

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-30 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
amount of bleeding during operation | 0 minute - 180 minute
  total amount of bleeding during surgery
operation duration time | 0 minute - 180 minute
  time between initial and end of the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Alku Alanya Education and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided